CLINICAL TRIAL: NCT04234126
Title: Does the Gallbladder Status Influence the Occurence of Post-Endoscopic Retrograde Choledochopancreatography(ERCP) -Choledocholithiasis
Brief Title: The Relationship Between Post-ERCP-choledocholithiasis and Gallbladder Status
Status: Completed | Type: Observational
Sponsor: Hepatopancreatobiliary Surgery Institute of Gansu Province (Other)
Responsible Party: Principal Investigator, Wenbo Meng, M.D., Ph. D, Director of surgery, Hepatopancreatobiliary Surgery Institute of Gansu Province
Other Study IDs: Gallbladder status and PEC
Record Dates: First submitted 2020-01-13; First posted 2020-01-21 (Actual); Last update posted 2021-11-19 (Actual); Status verified 2021-11

CONDITIONS: Cholecystitis
Keywords: ERCP; Acute purulent cholecystitis; Bile duct stone; PEC(post-ERCP-choledocholithiasis)
MeSH Terms: conditions — Cholecystitis; Cholecystolithiasis | interventions — Cholangiopancreatography, Endoscopic Retrograde

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: ERCP — Routine ERCP for CBD stone with the gallbladder in situ, the chronic gallbladder status was defined as gallbladder wall thickness≥4mm, chronic cholecystitis, polyps,crudely or calculus .

SUMMARY:
In this retrospective study, the investigators evaluate the relationship of post-ERCP-choledocholithiasis(PEC ) and the gallbladder status as a risk factor.

DETAILED DESCRIPTION:
When patients have common bile duct(CBD) stones, ERCP is widely used for stone extraction instead of clinical operation. ERCP has many advantages like less injury or faster recovery. However, according to literature, ERCP will has a mostly 10% possibility to get an acute purulent cholecystitis, which often requires emergency intervention, therefore, it is necessary to know if the gallbladder status(chronic disease) is one of the important risk factors of PEC like the gallbladder wall thickness, chronic cholecystitis, polyps,crudely or calculus.

.

ELIGIBILITY:
Inclusion Criteria:

* Routine ERCP for CBD stone patients with gallbladder in situ

Exclusion Criteria:

* Unwillingness or inability to consent for the study
* Unstable vital signs Coagulation dysfunction (INR>1.5) and low peripheral blood platelet count (<50×10 ^9 / L) or using anti-coagulation drugs
* Any Prior surgery for CBD including ERCP
* Preoperative coexistent diseases: acute pancreatitis, GI tract hemorrhage, severe liver disease (such as decompensated liver cirrhosis, liver failure and so on), septic shock
* Biliary- duodenal fistula confirmed during ERCP
* Pregnant women or breastfeeding

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Routine ERCP patients with CBD stones
Sampling Method: Probability Sample
Enrollment: 1117 (Actual)
Dates: Start 2020-01-31 (Actual); Primary Completion 2021-11-18 (Actual); Study Completion 2021-11-18 (Actual)

PRIMARY OUTCOMES:
Number of Acute PEC(post-ERCP-cholecystitis ) | 1 month
  When the PEC occurs, the temperature should be more than 38 celsius degree, right upper abdominal pain, the total amount of the White Blood Cell (WBC) is above normal for the patients who with the gallbladder wall thickness under ultrasound examination.

SECONDARY OUTCOMES:
Number of Participants with Pancreatitis | 1 month
  Typical abdominal pain, with the level of serum amylase increasing at least 3 times of the normal range within 24 hours after ERCP.
Number of Participants with Cholangitis | 1 month
  Temperature should be more than 38 celsius degree, chills, with right upper abdominal pain, blood routine showing the total amount of the White Blood Cell (WBC), and the amount of polymorphonuclear neutrophil(PMN) are above normal
Number of Participants with Perforation | 1 month
  Typical abdominal pain,abdominal muscle tension, and there are also radiographic evidence suggesting
Number of Participants with bile duct stents | 1 month
  If it is necessary to get the patients drainage, Number of Participants with stents or endoscopic nasobiliary drainage (ENBD) should be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Wenbo Meng, M.D., Ph. D., Principal Investigator — Hepatopancreatobiliary Surgery Institute of Gansu Province
Locations (1):
- Hepatopancreatobiliary Surgery Institute of Gansu Province, Lanzhou, Gansu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cao J, Ding X, Wu H, Shen Y, Zheng R, Peng C, Wang L, Zou X. Classification of the cystic duct patterns and endoscopic transpapillary cannulation of the gallbladder to prevent post-ERCP cholecystitis. BMC Gastroenterol. 2019 Aug 5;19(1):139. doi: 10.1186/s12876-019-1053-6. PMID 31382888
- [Derived] Jin B, Wang Y, Zhang X, Zhao J, He W, Jin K, Liu Z, Zhong R, Ma Y, Dong C, Lin Y, Zhu X, Zhu K, Zhang L, Yue P, Li S, Yuan J, Li X, Meng W. Identifying high-risk patients having ERCP as a day surgery with an online prediction platform: Multicohort validation of a machine learning model. Endosc Int Open. 2025 Dec 16;13:a27331387. doi: 10.1055/a-2733-1387. eCollection 2025. PMID 41567602
- [Derived] Zhang X, Yue P, Zhang J, Yang M, Chen J, Zhang B, Luo W, Wang M, Da Z, Lin Y, Zhou W, Zhang L, Zhu K, Ren Y, Yang L, Li S, Yuan J, Meng W, Leung JW, Li X. A novel machine learning model and a public online prediction platform for prediction of post-ERCP-cholecystitis (PEC). EClinicalMedicine. 2022 May 13;48:101431. doi: 10.1016/j.eclinm.2022.101431. eCollection 2022 Jun. PMID 35706483